CLINICAL TRIAL: NCT04960735
Title: Value-based Healthcare for Outcomes in Breast and Lung Cancer in Europe
Brief Title: Implementation, Effectiveness and Impact of a Value Based Intervention for Patients with Breast or Lung Cancer
Acronym: VOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosistemak Institute for Health Systems Research (Other)
Collaborators: Hospital de Cruces (Other); Hospital Donostia (Other); Hospital Universitario 12 de Octubre (Other); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other); Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other); Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other); Onze Lieve Vrouwziekenhuis Aalst (Other); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: INT/2020/VOICE
Record Dates: First submitted 2021-06-11; First posted 2021-07-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Lung Cancer
Keywords: Value-Based Healthcare; Breast Cancer; Lung Cancer; Patient Health Outcomes; Patient's perspective; Patient Reported Outcomes Measures (PROMs); Patient Reported Experience Measures (PREMs); Patient quality of life; Healthcare process; Cost analyses
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A single group intervention that will collect health-related Quality of Life evidence from patients with cancer from 13 hospitals for six months. The multicentre study combines an implementation research component and effectiveness, using quantitative and qualitative methods for data collection and analysis. Outcomes will be analysed not only at individual level but also at health organisation level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with cancer (patients with breast cancer and patients with lung cancer) (Experimental): Health-related Quality of Life evidence was collected from patients with cancer (patients with breast cancer and patients with lung cancer) for six months. The evidence was collected by means of health related and patient reported questionnaires (ICHOM standard sets for breast cancer and lung cancer).
  Patients were monitored for six months. Intervention outcomes were monitored at different times: for patients with breast cancer, at the start (on recruitment which coincided with diagnosis) and at six months; for patients with lung cancer, at the start (on recruitment which coincided with diagnosis), at three and at six months.
  Interventions: Other: VOICE intervention

INTERVENTIONS:
Other: VOICE intervention — The intervention consists of four stages:
  * S1, Value identification and description of current care processes: Needs are detected from two perspectives: feedback from patients and mapping of healthcare processes. ICHOM questionnaires are reviewed. Patient surveys and clinical forms are developed. The methodology for cost analysis is set up.
  * S2, Intervention implementation: Patients are recruited according to the eligibility criteria. Their care follows the current healthcare pathway and information is collected at different time points.
  * S3, Assessment of outcomes and continued benchmarking: Data and costs are analysed at both local level and Community level (benchmarking). Interviews and focus groups are held (optional). Root cause analysis is performed.
  * S4, Best practice sharing: Identifying what lessons could be learned from the best-performing sites, according to the results of the VOICE community benchmarking and following qualitative techniques.

SUMMARY:
VOICE project aims to guide health services in their reorganization towards the provision of the highest value care for the patient at the best cost. VOICE is targeted to patients with breast and lung cancer. The purpose is to offer a new innovative strategic framework based on value-based healthcare model to these patients in Europe. VOICE Community consists of 13 hospitals across Europe working collaboratively to implement this approach.

The Community addresses what matters most to patients by measuring patient reported health outcomes in routine clinical practice on a systematic and long-term basis, by including patients´ perspective in clinical decision-making, improving patient empowerment and physician-patient communication, assessing the impact on costs of the processes implemented, identifying factors for a successful implementation of value-based healthcare and boosting knowledge generation and best practice exchange across Europe.

The VOICE ambition is to collect the health-related Quality of Life evidence from more than 1000 patients (patients with breast cancer and patients with lung cancer), by means of health related and patient reported questionnaires (ICHOM, International Consortium for Health Outcome Measurements, standard sets). Hospitals will go further by assessing the satisfaction, acceptability, relationship with professionals or decision-making process with patients.

The VOICE Community will benchmark health outcomes and related costs to improve care delivery of these patients.

DETAILED DESCRIPTION:
VOICE is a Europe-wide Hospital Community pioneering in the assessment of value-based healthcare outcomes related to breast and lung cancer. The VOICE Community members have extended experience in value-based healthcare paradigm as they founded the community in 2018 in continuity with in the All.Can initiative launched by International Consortium for Health Outcome Measurements (ICHOM).

VOICE aims to implement the innovative value based healthcare approach for patients with breast cancer or lung cancer in routine practice to transform care provision and place the patient at the centre of the system. The project will assess the implementation process, the effectiveness of clinical practice and its impact on costs grouped by process for an intervention-based measurement of outcome values for patients with breast or lung cancer. As a result is expected to (i) analyse the effectiveness of an intervention based on measuring outcome values for patients in order to improve patient empowerment, shared decision-making, and physician-patient communication; (ii) assess the impact of an intervention based on measuring outcome values for patients on costs grouped by clinical process, and in the organisation of healthcare by processes and (iii) integrate the measurement of value-based health outcomes in everyday clinical practice for organisations both systematically and long term.

This study duration will be three years and a half.

* Preparation period (July-December 2018): the intervention was defined; the data battery to be collected was designed; the systems required for that purpose were developed; and professionals participating in the study were recruited and trained.
* Intervention period (January 2019-June 2020): all processes set forth were activated; patient recruitment and follow-up, as well as data collection started.
* Analysis and benchmarking period (June 2020-June 2023): data collected will be analysed and outcomes will be compared among organisations participating in the study and corresponding dissemination.

More than 1,000 patients were progressively recruited in 13 pilot sites (European Hospitals) when diagnosed with breast or lung cancer. Patients who met the eligibility criteria described below were invited to take part in the study once diagnosed at the hospital. Medical professionals (gynaecology, oncology, pneumology and thoracic surgery consultants) explained the study and provided the patients with the information sheet and informed consent form.

Recruitment was conducted in the first six months and patients were monitored for at least six months or until death, if that occurred first. Intervention outcomes were monitored at different times: at the start (on recruitment which coincided with diagnosis); at 6 months in breast cancer; and at the start (on recruitment which coincided with diagnosis), at 3 months; and after 6 months in lung cancer.

This multicentre prospective study combines an implementation research component and an effectiveness component, using quantitative and qualitative methods for data collection and analysis. Quantitative analysis includes a descriptive analysis of all variables included in the study. Categorical variables will be shown using frequencies and percentages, n (%). Continuous variables with normal distribution will be shown as standard deviation (SD). Continuous variables with non-normal distribution will be shown as median and first and third quartiles (Q1, Q3). Pre and post intervention differences between categorical variables will be calculated with McNemar's test used on paired data. In continuous variables, the Student´s t test will be used on paired data; or the Wilcoxon rank sum test for variables with normal and non-normal distributions, respectively. Moreover, regression models for the pre/post difference will be proposed to assess whether that difference varies from 0. Models will be adjusted by possible determinant factors such as gender and other socio-demographic elements.

The qualitative analysis to be carried out at the end of the intervention will include semi-structured interviews and focus groups methods. Analyses will be performed at individual level (patient) and at organisational level (costs).

Data management will meet the current European Union (EU) General Data Protection Regulations (GDPR) and shall include detailed information on the procedures in terms of data collection, conservation, protection, reuse and/or destruction. The project will only obtain essential data, and will never share patients' personal data or raw anonymous data. Data obtained will be used for assessment purposes, impact valuation and to increase the empirical base. Templates are based on ICHOM data dictionary for breast cancer and lung cancer where each variable is coded and responses are typified.

VOICE will follow the procedures indicated in the new general data protection regulation No 2016/679 that has been recently applied in Europe for the data access, protection and sharing.

The Community partners have signed an agreement to access and to share data.

ELIGIBILITY:
Inclusion Criteria for patients with breast cancer:

* male and female over 18
* recently diagnosed with invasive stage I-IV cancer, or Ductal Carcinoma in Situ (DCIS)
* undergoing any treatment type (surgery, radiotherapy, chemotherapy, hormone therapy and/or targeted therapy).

Inclusion Criteria for patients with lung cancer:

* male and female over 18
* newly diagnosed with lung cancer
* eligible to receive curative or palliative care treatment.

Exclusion Criteria for patients with breast cancer:

* With rare tumours
* With Lobular Carcinoma In Situ (LCIS)
* With recurring illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline overall well-being for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.. Lung Cancer patients completed the PROMs questionnaires at baseline, and after three and six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Asthenia and fatigue (including physical functioning) at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Emotional functioning (also including anxiety and depression) for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Cognitive functioning for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Social and working functioning (also including financial impact) for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Body image for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC QLQ---BR23 (BR23: Breast Cancer Module).
Change from baseline Sexual functioning for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC QLQ---BR23 (BR23: Breast Cancer Module).
Change from baseline Satisfaction with breasts for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire BREAST---Q ---Satisfaction with Breast (The BREAST-Q © is a multiscale, multimodule, patient-reported outcome instrument (PRO) measuring health-related quality of life and patient satisfaction in women who undergo breast surgery.Domain Patient satisfaction: Satisfaction with breasts).
Change from baseline Arm and breast symptoms for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC QLQ---BR23 (BR23: Breast Cancer Module).
Change from baseline Adverse effects: vasomotor symptoms for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC QLQ---BR23 (BR23: Breast Cancer Module).
Change from baseline Adverse effects: peripheral neuropathy for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC QLQ---LMC21 (questionnaire for assessment of patient-reported outcomes during treatment of colorectal liver metastases) -- single item.
Change from baseline Adverse effects: Arthralgia for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaires EORTC QLQ---BR23, EORTC QLQ---LMC21 -- (questionnaire for assessment of patient-reported outcomes during treatment of colorectal liver metastases) single item and FACT (Functional Assessment of Cancer Therapy) -- ES (Endocrine Subscale) (single item).
Change from baseline Vaginal symptoms for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire FACT (Functional Assessment of Cancer Therapy) -- ES (Endocrine Subscale) (single item).
Change from baseline Quality of life for patients with breast cancer at 6 months | Breast Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the standardised measure EQ-5D (5D: Dimensions) (EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys) for the measurement of health-related quality of life. EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. On the scale, a value of 100 indicates the best imaginable state of health while a value of 0 the worst imaginable state of health.
Change from baseline Global health status / Quality of life for patients with Lung Cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Fatigue for patients with lung cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Social function for patients with lung cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Physical functioning for patients with Lung Cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Emotional functioning for patients with lung cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Cognitive function for patients with Lung Cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with breast cancer by means of completion of the questionnaire EORTC (European Organization for Research and Treatment of Cancer) QLQ (quality of life questionnaire) -- C30.
Change from baseline Pain for patients with lung cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with lung cancer by means of completion of the questionnaires EORTC QLQ---C30 and EORT QLQ-LC13 (a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials).
Change from baseline Shortness of breath for patients with Lung Cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with lung cancer by means of completion of the questionnaire EORT QLQ-LC13 (a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials).
Change from baseline Cough for patients with lung cancer at 6 months | Lung Cancer patients completed the PROMs questionnaires at baseline and after six months.
  Outcome measure reported by patients with lung cancer by means of completion of the questionnaire EORT QLQ-LC13 (a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials).

SECONDARY OUTCOMES:
Rate of survival of patients with Breast Cancer | For Breast cancer patients, during the intervention: at baseline and at six months.
  Percentage of patients alive after completion of the study For Lung Cancer: Overall survival, Cause of death, Quality of death.
Rate of survival of patients with Lung Cancer | For Breast cancer patients, during the intervention: at baseline, and at three and at six months.
  Percentage of patients alive after completion of the study
Number of patients suffering serious treatment-related complications due to care of treatment for breast cancer | For Breast cancer patients, during the intervention: at six months since the diagnostic.
  For Breast Cancer: Number of patients with serious treatment-related complications defined as death, life-threatening, requiring in-patient hospitalization or prolongation of existing hospitalization, resulting in persistent or significant disability or incapacity, or a congenital anomaly/birth effect / Total number of patients
Number of patients suffering serious treatment-related complications due to care of treatment for lung cancer | For Lung Cancer patients, during the intervention: at six months since the diagnostic.
  For Lung Cancer: Number of patients with serious treatment-related complications defined as death, life-threatening, requiring in-patient hospitalization or prolongation of existing hospitalization, resulting in persistent or significant disability or incapacity, or a congenital anomaly/birth effect / Total number of patients
Average total cost per patient with breast cancer | For Breast cancer patients, during the intervention at 12 months period since the diagnostic
  Sum of costs associated to the resource use of the total number of patients / Total number of patients
Average total cost per patient with lung cancer | For Lung cancer patients, during the intervention at 12 months period since the diagnostic
  Sum of costs associated to the resource use of the total number of patients / Total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Ane Fullaondo, Ph.D., Study Chair — Biosistemak (formerly Kronikgune)
Locations (8):
- Olv Aalst, Aalst, Flanders, Belgium
- Institut de Cancerologie de l'Ouest, Angers, Maine Et Loira, France
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forlì-Cesena, Italy
- Instituto Português de Oncologia do Porto, Porto, Portugal
- Spain (4):
  - Donostia University Hospital, San Sebastián, Gipuzkoa
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - 12 Octubre University Hospital, Madrid, Madrid
  - Cruces University Hospital, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Lorenzo B, Gorostiza A, Alayo I, Castelo Zas S, Cobos Baena P, Gallego Camina I, Izaguirre Narbaiza B, Mallabiabarrena G, Ustarroz-Aguirre I, Rigabert A, Balzi W, Maltoni R, Massa I, Alvarez Lopez I, Arevalo Lobera S, Esteban M, Fernandez Calleja M, Gomez Mediavilla J, Fernandez M, Del Oro Hitar M, Ortega Torres MDC, Sanz Ferrandez MC, Manso Sanchez L, Serrano Balazote P, Varela Rodriguez C, Campone M, Le Lann S, Vercauter P, Tournoy K, Borges M, Oliveira AS, Soares M, Fullaondo A; VOICE Study Group. European value-based healthcare benchmarking: moving from theory to practice. Eur J Public Health. 2024 Feb 5;34(1):44-51. doi: 10.1093/eurpub/ckad181. PMID 37875008
- [Background] Garcia-Lorenzo B, Alayo I, Arrospide A, Gorostiza A, Fullaondo A; VOICE Study Group. Disentangling the value equation: a step forward in value-based healthcare. Eur J Public Health. 2024 Aug 1;34(4):632-638. doi: 10.1093/eurpub/ckae060. PMID 38878265
- See also: Description of VOICE project in the web page of the Sponsor — https://www.kronikgune.org/en/european-community-voice/